CLINICAL TRIAL: NCT01661127
Title: Phase 0 Clinical Study of PET/CT and Association With Metabolic Syndrome/Depressive Symptoms in Psoriasis
Brief Title: Clinical Study of PET/CT and Association With Metabolic Syndrome/Depressive Symptoms in Psoriasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PNUHDM-psoriasis
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Psoriasis; Metabolic Syndrome; Depression
MeSH Terms: conditions — Psoriasis; Metabolic Syndrome; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood and 18-F-FDG PET/CT images
Oversight: Data Monitoring Committee: No

SUMMARY:
Psoriasis is associated with increases in markers of inflammation in the skin and blood and increasingly is thought to be a systemic inflammatory disease and risk factor for incident diabetes mellitus, myocardial infarction, stroke, and premature cardiovascular death. Furthermore, it is important for clinicians to be aware that psoriasis can have a substantial emotional impact on an individual, which is not necessarily related to the extent of skin disease.

FDG-PET/CT represents an innovative approach to studying systemic inflammation in a manner that is sensitive, quantifiable, and anatomically localizable. Also, recent study show that chronic disease such as end stage renal disease with depressive symptoms have decreased cerebral glucose metabolism in several brain areas in F-18-FDG PET/CT. So this protocol was designed to evaluate usefulness of PET/CT to detect systemic inflammation and abnormality of cerebral glucose metabolism and association with metabolic syndrome/major depressive symptoms in patients with psoriasis.

DETAILED DESCRIPTION:
10 Patients with psoriasis

1. Evaluate PASI score
2. Evaluate comorbidity with metabolic syndrome

   * Body mass index(BMI)
   * Checking blood pressure
   * Checking blood sugar
   * Smoking and drinking history
   * Checking blood cholesterol level
   * Risk factors of cardiovascular disease
3. PET/CT for measuring the extent and site of psoriasis with inflammation

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of plaque type psoriasis
* at least 18 years old

Exclusion Criteria:

* those who cannot understand questionnaire
* those who take antidepressant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of diagnosed with psoriasis in Pusan National University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Beck depression inventory scoring and Korean Hamilton depression scale scoring | Day 0 and 28 weeks later

SECONDARY OUTCOMES:
Brain glucose uptake using PET/CT | Day 0 and 28 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Soo Kim, Ph D., Study Chair — Pusan National University Hospital
Locations (1):
- Department of dermatology, Pusan National University Hospital, Busan, Busan, South Korea